CLINICAL TRIAL: NCT05060081
Title: Comparison of Pilates and Traditional Plank on Core Muscle Strength, Balance and Agility in Recreational Badminton Players
Brief Title: Comparison of Pilates and Traditional Plank in Recreational Badminton Players.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01019 Najla Ammar
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Sports Physical Therapy
Keywords: Sports Rehabilitation; Pilates; Planks; Strength; Balance; Agility; Badminton

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates exercise program group (Experimental): Pilates exercise program group will perform five exercises.
  Interventions: Other: Pilates exercise program group
- Traditional plank exercise program group (Active Comparator): Traditional plank exercise program group will perform five exercises.
  Interventions: Other: Traditional plank exercise program group

INTERVENTIONS:
Other: Pilates exercise program group — Pilates exercise program group will do a warm-up for 10 minutes and then perform five exercises includes standing footwork, hundreds with knee straight, articulating bridge, rolling like a ball, plank for 25 minutes. For first three weeks, each player will do 8 repetitions × 3 sets of exercises and for next three weeks, each player will do 15 repetitions × 3 sets of exercises. There will be cool-down for 10 minutes after exercises. Total program will be of 45 minutes.
  Arms: Pilates exercise program group
Other: Traditional plank exercise program group — Traditional plank exercise program group will do a warm-up for 10 minutes and then perform five exercises includes prone bridge, side bridge, supine bridge on exercise ball, prone bridge on exercise ball, superman on exercise ball. For first three weeks, each player will do 8 repetitions × 3 sets of exercises and for next three weeks, each player will do 15 repetitions × 3 sets of exercises. There will be cool-down for 10 minutes after exercises. Total program will be of 45 minutes.
  Arms: Traditional plank exercise program group

SUMMARY:
To compare the effects of Pilates exercise and traditional plank exercise training on core muscle strength, balance and agility in recreational badminton players

DETAILED DESCRIPTION:
In modern era, badminton is one of the most famous and played sports worldwide. As compared to other indoor games, badminton is considered to be the finest sports as it occupies a place of pride for both as an individual and team sport. It is a technical and complex sport activity that need massive core strength and whole body strength in strokes, powerful smashes, alertness, well balance and coordination during postural movement in the premises of the court. Notable, to be competitive in badminton, players need to be able to move quickly toward well balanced position that permits them to tackle quickly to hit the shuttlecock.

The purpose of this study is to compare the effects of pilates exercises and traditional plank exercise training on core muscle strength, balance and agility in recreational badminton players.

ELIGIBILITY:
Inclusion Criteria:

* Players playing badminton for > 1 year
* Players engaging in badminton ≥ 3 days in a week

Exclusion Criteria:

* History of any injury in past 6 months
* Those players having musculoskeletal, neurological or cardiorespiratory problems
* Those players who have any medical conditions

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Star Excursion Balance Test (SEBT) | Six weeks
  The SEBT was performed with the player standing at the center of a grid placed on the floor, with 8 lines extending at 458 increments from the center of the grid. The 8 lines were labeled according to the direction of excursion relative to the stance leg: Antero-lateral (AL), Anterior (A), Antero-medial (AM), Medial (M), Poster-medial (PM), Posterior (P), Poster-lateral (PL), and Lateral (L). To perform the SEBTs, the player maintained a single-leg stance while reaching with the opposite leg as far as possible. The player lightly touched the farthest point possible on the line with the most distal part of the reach foot then returning to a bilateral stance while maintaining their balance. The distance was measured from the center of the grid to the touch point with a tape measure in centimeters. There will be two assessments, at baseline before the start of exercise program and at the end of six weeks intervention.
One Min Sit Up Test | Six weeks
  Core muscles Strength was measured by one min Sit up test and Prone Bridge Test (Plank Test).The subject lay supine on the floor with 90° flexion in the knee joints, hands at the side of their head, and with elbows pointing straight forward. To do a correct sit-up execution the elbows should touch the knees and then go back so the shoulders touch the floor. The number of repetitions performed was recorded. There will be two assessments, at baseline before the start of exercise program and at the end of six weeks intervention.
Badcamp Agility Test | Six weeks
  The Badcamp Agility test was performed with players standing at the middle of the badminton court. Six targets were placed at six ends of the court. The players were give warning signal and the examiner started marking the corners which players have to follow. The players have to touch all 6 markers as marked by the examiner in an undecided manner. Each participant performed the test 3 times, and the shortest time was considered for analysis. At least 1 minute of rest was given between trials. There will be two assessments, at baseline before the start of exercise program and at the end of six weeks intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Aadil Omer, Ph.D.*, Principal Investigator — Riphah International University
Locations (1):
- Sports Complex, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No